CLINICAL TRIAL: NCT00774501
Title: A Pilot Study to Assess the Feasibility of Using Anesthesia and Suspended Ventilation to Immobilize Liver Tumors During Radiotherapy
Brief Title: The Feasibility of Using Anesthesia and Suspended Ventilation to Immobilize Liver Tumors During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-117
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cancer
Keywords: Anesthesia; suspended ventilation
MeSH Terms: conditions — Liver Neoplasms | interventions — Anesthesia, General

ARMS (1):
- treatment of metastatic liver disease (Experimental): The intervention is the use of image guidance with general anesthesia and suspended ventilation during treatment delivery. This will allow precise localization and delivery of dose to the tumor.
  Interventions: Procedure: image guidance with general anesthesia and suspended ventilation during treatment delivery

INTERVENTIONS:
Procedure: image guidance with general anesthesia and suspended ventilation during treatment delivery — All study patients will undergo marker implantation approximately 2 weeks prior to the PET-CT simulation and treatment planning. PET-CT is performed for treatment planning purposes. This part of the process is in routine clinical use at MSKCC.
  Three cone beam imaging scans and an IV contrast injection just prior to the first cone beam scan will be added to the standard procedure. The use of these two techniques is investigational.
  The treatment delivery will make use of general anesthesia and suspension of mechanical ventilation to render the patient apneic during both target localization and dose delivery. This will allow the dose to be delivered more precisely than the techniques currently in use, thus allowing the use of smaller treatment margins and reducing the high dose exposure of healthy liver tissue. These measures have not previously been used for treatment delivery.

SUMMARY:
Liver tumors are hard to treat with radiation because the liver moves every time you breathe. The purpose of this study is to test a new and possibly more accurate way of treating liver tumors. When a person is asleep under anesthesia, it is safe to stop breathing motion for a while. The liver will stop moving and radiation can be given to a liver tumor. The study is being done to see if radiation can be given to liver tumors safely and accurately in this way.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible to receive external beam intensity modulated radiotherapy for liver cancer
* Age:21<80
* KPS > or = to 80
* Able to tolerate immobilization cradle positioning
* Able to give informed consent
* Histologically confirmed diagnosis of solid tumor malignancy
* Liver metastases visualized on CT imaging (obtained within approximately 6 months from enrollment).
* Target lesion ≤ or = to 8 cm in maximal diameter
* In the case of multiple liver metastases, only one lesion will be targeted per treatment session. Typically the target lesion will be the lesion which is progressing or the cause of symptoms. The target lesion will be picked in consultation with the referring physician.

Exclusion Criteria:

* Lymphoid primary histology (lymphoma/leukemia)
* Single metastasis in an operable patient. Operable lesions will only be considered for enrollment in the protocol if the patient refuses resection of the metastasis.
* Target lesion > 8 cm in maximal diameter
* Cirrhosis of the liver (Child's C)
* Liver function enzymes (AST, ALT) > 3x normal , obtained within 1 month of treatment.
* < 500 cc uninvolved liver
* Unable to tolerate intravenous CT contrast
* Serum Hemoglobin < 9.0 (obtained within 1 month of treatment)
* Presence of untreated brain metastases
* Severe pulmonary disease (O2 dependent, unable to walk a flight of stairs)
* Unstable cardiac status
* Unstable angina
* Significant abnormal 12 lead EKG (non sinus arrhythmia or ischemia unsuitable for general anesthesia)
* Congestive Heart Failure
* Abnormal kidney function (serum creatinine > 1.5) obtained within 1 month of treatment
* Platelet count <70.000. (obtained within 1 month of treatment).
* INR > 2.0 (obtained within 1 month of treatment)
* Marker seed placement not possible
* Implanted defibrillator/pacemaker
* Evidence of increased intracranial pressure
* Significant ascites
* Morbid Obesity
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess safety & feasibility of single dose image-guided intensity modulated radio (IG-IMRT) using gen anesthesia with apneic oxygenation & controlled ventilation to temp suspend respiratory motion for tx of mets liver disease during localization & tx. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org